CLINICAL TRIAL: NCT04539080
Title: Heart Rate Variability and Electroencephalography Analysis in Laparoscopic Surgery With or Without Transversus Abdominis Plane Block
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20MMHIS210e
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Autonomic Nervous System; Nerve Block; Laparoscopy; Anesthesia and Analgesia; EEG
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-operative transversus abdominis plane block: The group with transversus abdominis plane block before laparoscopic surgeries with a standard pain control protocol
  Interventions: Procedure: transversus abdominis plane block
- Traditional pain control group: The group with a standard pain control protocol

INTERVENTIONS:
Procedure: transversus abdominis plane block — transversus abdominis plane block group
  Groups: Pre-operative transversus abdominis plane block

SUMMARY:
Heart rate variability(HRV) and electroencephalography(EEG) has been used widely in anesthetic practice nowadays. One of the most dominant applications is the nociception-analgesia balance. Some evidence support that heart rate variability correlates with perioperative stimulation and postoperative pain score. There are some new evidence support EEG correlated with anesthesia depth and analgesic balance. However, the heterogeneity between the studies and interference factors has limited their usage in clinical practice. On the other hand, peripheral nerve block is broadly used as a routine technique with general anesthesia, but few studies discuss the effect on heart rate variability. Our study focuses on the different HRV and EEG patterns of incision and insufflation during laparoscopic surgery with general anesthesia. Furthermore, we measure the effect of transversus abdominis plane nerve block to heart rate variability during surgery. By this comparison, we can discuss the influences of somatic stimulation, visceral stimulation, and pneumoperitoneum to heart rate variability, and then improve the accuracy of HRV-based nociception-analgesia monitors.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years of age male or female
* American Society of Anesthesiologists (ASA) physical status classification I or II
* capacity to give informed consent

Exclusion Criteria:

* major cardiovascular and cerebral vascular disease, arrhythmia, respiratory disease, diabetes mellitus with evidence of neuropathy; ASA physical status classification III or greater; a documented or self-reported history of chronic pain; acute or chronic opioid analgesic use; dysautonomia; and intraoperative muscarinic anticholinergic administration during the time of monitoring.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: scheduled to undergo general anesthesia for laparoscopic surgery (cholecystectomy or appendectomy) at Taitung MacKay memorial hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Different heart rate variability pattern during laparoscopy | 6 months
  Different heart rate variability pattern in incision and inflation with or without TAP block

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Chun Wang, MD, Principal Investigator — Taitung Mackay Memorial Hospital
Locations (1):
- Taitung MacKay memorial hospital, Taitung, Taitung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang TC, Li WY, Lai JC, Kuo TBJ, Yang CCH. Nociception Effect on Frontal Electroencephalogram Waveform and Phase-Amplitude Coupling in Laparoscopic Surgery. Anesth Analg. 2024 May 1;138(5):1070-1080. doi: 10.1213/ANE.0000000000006609. Epub 2023 Jul 10. PMID 37428681